| STATISTISKA KONSULTGRUPPEN | Statistica | ıl Analysis Plan |
|---|---|---|
| Protocol: Clinical performance of a new implant system for bone CBAS553 | | |
| conduction hearing | Version: 1.0 | |

# Statistical Analysis Plan

ATB System

**CBAS5539** 

Clinical performance of a new implant system for bone conduction hearing

Open, prospective, multicentre clinical investigation. 3-month investigation with an additional 9 months of follow-up

2018-04-16

NCT0386135

# STATISTISKA KONSULTGRUPPEN Protocol: Clinical performance of a new implant system for bone conduction hearing Protocol No: CBAS5539 Version: 1.0 

# **Table of Contents**

| 1 | | etails | |
|---|---|---|---|
| | | dy Objectives | |
| | | dy Design | |
| | | vchart | |
| | | rice/Treatment Groups | |
| | | nple Size | |
| | 1.5.1 | Sample size calculation for the primary efficacy analysis: | |
| | 1.5.2 | Sample size estimation for the primary safety analysis at 6 months | |
| | 1.5.3 | Overall sample size considerations | |
| 2 | | opulations | |
| | | inition of Study Populations | |
| | 2.1.1 | Intent-to-Treat Population (Full Analysis Set) | |
| | 2.1.2 | Per-Protocol Population | |
| | 2.1.3 | Safety Population | |
| 3 | | ariables | |
| | | eline variables | |
| | 3.1.1 | Demographics | |
| | 3.1.2 | Baseline Characteristics | |
| | 3.1.3 | Medical and Surgical History | |
| | 3.1.4 | Prior and Concomitant Medications | |
| | 3.1.5 | Concomitant Treatments/Procedures | |
| | | cacy Variables/endpoints | |
| | 3.2.1 | Primary Efficacy Variables/endpoints | |
| | 3.2.2 | Secondary Efficacy Variables/endpoints | |
| | | ety Variables/Endpoints | 12 |
| | 3.3.1 | Implant site evaluation | |
| | 3.3.2 | Adverse Events | |
| | 3.3.3 | Device deficiency | |
| | 3.3.4 | Audiogram | |
| 4 | | al Methodology | |
| | | neral Methodology | |
| | | ing of analyses | |
| | | ent Disposition and Data Sets Analysed | |
| | | tocol Deviations | |
| | | nographics and Baseline Characteristics | |
| | | operation variables | |
| | | dical and Surgical History | |
| | | or and Concomitant Medications | |
| | | ncomitant Treatments/Procedures | 15 |
| | | fficacy Analyses | |
| | 4.10.1 | Primary Efficacy Analysis | |
| | 4.10.2 | Secondary Efficacy Analyses | |
| | 4.10.3 | Tertiary Efficacy Analyses | |
| | | afety Analyses | |
| | 4.11.1 | Implant site evaluation | |
| | 4.11.2 | Adverse Events | |
| | 4.11.3 | Device deficiency | |
| | 4.11.4 | Audiogram | |
| _ | | andling of change in Osia version of Fitting Software | |
| 5 | | Analyses | |
| 6 | | s of Analysis from Protocol | |
| 7 | | f Table, Figures and Listings | |
| | | ing of Tables | |
| | 7.2 Listi | ing of Figures | 21 |

| Protocol: Clinical performance of a new implant system for bone conduction hearing | Protocol No: CBAS5539 | |
|---|---|---|
| | Version: 1.0 | Page 3 of 2 |
| 7.3 Listing of Listings | | |

| STATISTISKA KONSULTGRUPPEN | Statistica | l Analysis Plan |
|---|---|---|
| Protocol: Clinical performance of a new implant system for bone | Protocol No:<br>CBAS5539 | |

# **LIST OF ABBREVIATIONS**

| Abbreviation | Definition |
|---|---|
| ADE | Adverse Device Effect |
| AE | Adverse Event |
| AESI | Adverse events of special interest |
| APHAB | Abbreviated Profile of Hearing Aid Benefit |
| ATB | Active transcutaneous Baha |
| ATC | Anatomic Therapeutic Chemical classification system |
| BC | Bone Conduction |
| BFS | Baha Fitting Software |
| d | Day |
| dB | Decibel |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DD | Device Deficiency |
| HUI | Health Utilities Index |
| Hz | Hertz |
| ITT | Intention to treat |
| m | Month |
| Max | Maximum |
| min | Minute |
| Min | Minimum |
| mm | Millimetre |
| PP | Per protocol |
| PT | Preferred Term |
| PTA | Pure Tone Average |
| SADE | Serious Adverse Device Effect |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SEM | Standard Error of the Mean |
| SOC | System Organ Class |
| SP | Sound Processor |
| SPM | Sound Processor Magnet |
| SSD | Single Sided Deafness |
| SSQ | The Speech, Spatial and Qualities of Hearing Scale |
| W | Week |
| WHO CC | World Health Organization Collaborating Centre for Drug Statistics Methodology |

| STATISTISKA KONSULTGRUPPEN | Statistica | l Analysis Plan |
|---|---|---|

# 1 STUDY DETAILS

# 1.1 Study Objectives

| Objectives and outcome measures | |
|---|---|
| Primary objective | Outcome measures/endpoints |
| To compare hearing performance with the Investigational device and the unaided hearing situation | Thresholds audiometry, free-field [PTA4,<br>Mean of 0.5, 1, 2 and 4 kHz]. Investigational<br>device (at 3 months) vs. Unaided. |
| | Adaptive speech in noise Matrix Test [speech-to-noise ratio, 50% speech understanding] (at 3 months). Investigational device vs. Unaided. |

| Secondary objectives | Outcome magazza landa cinta |
|---|---|
| To compare hearing performance with the Investigational device and the unaided hearing situation | Thresholds audiometry, free-field [PTA4, Mean of 0.5, 1, 2 and 4 kHz]. Investigational device (4 weeks, 6 and 12 months) vs. Unaided. |
| | Thresholds audiometry, free-field [0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0 and 8.0 kHz]. Investigational device vs. Unaided. |
| | Adaptive speech in noise Matrix Test<br>[speech-to-noise ratio, 50% speech<br>understanding]. Investigational device (6 and<br>12 months) vs. Unaided. |
| | Speech in quiet [% correctly perceived words<br>at 50dB, 65dB and 80dB SPL]. Investigational<br>device vs. Unaided. |
| | Feedback measurements. Investigational device. |
| To compare the self-reported assessments of hearing outcome with | Abbreviated Profile of Hearing Aid Benefit<br>(APHAB). Investigational device vs. Unaided. |
| the Investigational device and in a preoperative hearing situation | Health Utilities Index (HUI23S1EN.15Q). Investigational device vs. preoperative hearing situation |
| | Speech, Spatial and Qualities of Hearing<br>Scale (SSQ). Investigational device vs.<br>Unaided. |
| To collect surgical information | Soft tissue thickness |
| | Soft tissue reduction performed |
| | Type of anaesthesia |

| STATISTISKA KONSULTGRUPPEN | Statistica | l Analysis Plan |
|---|---|---|

| | <ul> <li>Surgery time</li> <li>Bone polishing/removal at the actuator site</li> <li>BI300 Implant length</li> <li>Location of BI300 Implant</li> <li>Surgical incision type/location</li> </ul> |
|---|---|
| To collect information about the magnet choice and daily use of sound processor | <ul> <li>Daily usage time</li> <li>Comfort</li> <li>Softpad use</li> <li>Choice of magnet strength</li> </ul> |
| To measure hearing performance preoperatively with a Baha BP110 Power Sound Processor on a Baha Softband | <ul> <li>Thresholds audiometry, free-field [PTA4, Mean of 0.5, 1, 2 and 4 kHz].</li> <li>Thresholds audiometry, free-field [0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0 and 8.0 kHz].</li> <li>Speech in quiet [% correctly perceived words at 50dB, 65dB and 80dB SPL]</li> <li>Adaptive speech in noise [speech-to-noise ratio, 50% speech understanding].</li> <li>BC Direct [0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0 and 6.0 kHz].</li> </ul> |

| Tertiary objective | Outcome measures/endpoints |
|---|---|
| To measure hearing performance preoperatively with a current hearing aid (if used by the patient) | <ul> <li>Adaptive speech in noise [speech-to-noise<br/>ratio, 50% speech understanding].</li> </ul> |

| Safety objectives | Outcome measures/endpoints |
|---|---|
| The primary safety analysis will be performed at 6 months | |
| Implant site evaluations | Numbness |
| Adverse Events and concomitant medication/treatment | Information will be collected from visit 2 and onwards. |
| Device deficiency | Information will be collected from Visit 2 and onwards. |
| Audiogram | Bone conduction thresholds preoperative and postoperative |

| STATISTISKA KONSULTGRUPPEN | Statistical Analysis Plan |
|---|---|
| Clinical performance of a new implant system for bone | w implant system for bone Protocol No: CBAS5539 |

# 1.2 Study Design

Open, prospective, multicentre clinical investigation. 3-month investigation (primary efficacy analysis) with an additional 9 months of follow-up. Primary safety analysis occurs during the investigation at 6 months.

| STATISTISKA KONSULTGRUPPEN | Statistical Analysis Plan |
|---|---|
| Clinical performance of a new implant system for bone | CBAS |

# 1.3 Flowchart

| | Visit 1 Pre- op testing | Visit 2<br>Surgery | Visit 3<br>Suture<br>removal | Visit 4 Fitting | Visit<br>5 | Visit<br>6 | Visit<br>7 | Visit<br>8 |
|---|---|---|---|---|---|---|---|---|
| Visit time point | | 0 | 2W | 4W | 6W | 3M | 6M | 12M |
| Visit window | | | ± 5D | ± 1W | ± 1W | ± 2W | ± 3W | ± 4W |
| Demographics | Х | | | | | | | |
| Medical history | Х | | | | | | | |
| Baseline characteristics | Х | | | | | | | |
| Audiogram | Х | | | | | X <sup>6</sup> | | X <sup>6</sup> |
| Eligibility criteria | Х | | | | | | | |
| Informed consent | Х | | | | | | | |
| Soft tissue thickness | Х | or X | | | | | | |
| Surgery <sup>1</sup> | | Х | | | | | | |
| IOTS | | Х | | | | | | |
| Suture removal | | | Х | | | | | |
| Sound processor fitting | X <sup>2</sup> | | | Х | Х | Х | Х | Х |
| Magnet choice | | | | Х | Х | Х | Х | Х |
| BC Direct | X <sup>2</sup> | | | Х | Х | Х | Х | Х |
| Feedback measurements | | | | Х | Х | Х | Х | Х |
| Free field thresholds | X <sup>2,3.4</sup> | | | Х | | Х | Х | Х |
| Speech recognition in quiet | X <sup>2,3, 4</sup> | | | х | | Х | Х | Х |
| Speech recognition in noise | X <sup>2,3, 4</sup> | | | х | | Х | Х | Х |
| APHAB | X <sup>3</sup> | | | | | Х | | Х |
| HUI | X <sup>4</sup> | | | | | Х | | Х |
| SSQ | X <sup>3</sup> | | | | | Х | | Х |
| Daily use <sup>5</sup> | | | | | Х | Х | Х | Х |
| Numbness | | | Х | Х | Х | Х | Х | Х |
| - · · · · · · | l | | | | l ,. | 1 ,. | | T |
| Device deficiency | | X | X | X | X | X | X | X |
| Adverse events | | Х | Х | Х | Х | Х | Х | Х |
| Concomitant medication/treatment | | Х | Х | Х | Х | Х | Х | Х |
| Extra visits as needed | | | | | | | | |

| STATISTISKA KONSULTGRUPPEN | Statistical Analysis Plan |
|---|---|
| Protocol: Clinical performance of a new implant system for bone | CBAS |

| | Visit 1 Pre- op testing | Visit 2<br>Surgery | Visit 3<br>Suture<br>removal | Visit 4 Fitting | Visit<br>5 | Visit<br>6 | Visit<br>7 | Visit<br>8 |
|---|---|---|---|---|---|---|---|---|
| Visit time point | | 0 | 2W | 4W | 6W | 3M | 6M | 12M |

<sup>&</sup>lt;sup>1</sup> Surgical variables: Soft tissue thickness (mm), Surgery time (time between first incision and last suture), Bone polishing/removal at the actuator site, Bl300 Implant length (4mm, 3 mm), Location of Bl300 Implant (mm), Type of anaesthesia (general, local), Soft tissue reduction performed (yes, no), Surgical incision type.

- <sup>2</sup> BahaPower Sound Processor (BP110) on Baha Softband
- <sup>3</sup> Unaided
- <sup>4</sup> In a preoperative hearing situation
- <sup>5</sup> Daily use: Usage time (hours/day), Comfort (visual analogue scale), Softpad use
- <sup>6</sup> Only bone conduction

# 1.4 Device/Treatment Groups

Only one device group is included in this study.

#### 1.5 Sample Size

#### 1.5.1 Sample size calculation for the primary efficacy analysis:

In order to achieve 90% power to detect a clinically significant difference of 10 dB in free-field hearing thresholds or 10 SNR between the unaided situation and the ATB System at the 3 months visit with Fisher's non-parametric permutation test for paired observations, one-sided test with significance level 0.025, on the ITT population 11 (PTA-4) and 13 (SNR) evaluable subjects are needed. The sample size was calculated using simulation on study id CBAS5675 (Cochlear 2017) data which used the simulated ATB system on Mixed/Conductive subjects. The within subject SD for change Unaided to ATB in PTA4 was 9.5 dB and 11.3 SNR. Since significant result want to be detected in both arms (SSD and Conductive/Mixed) 13+13=26 subjects should be included in the investigation.

#### 1.5.2 Sample size estimation for the primary safety analysis at 6 months

Primary safety analysis will be evaluated at 6 months and an estimation of 50 subjects results in 25 patient years at 6 months which will yield enough safety data for the primary safety analysis. At the 12 months analysis 50 subjects results in 50 patient years.

# 1.5.3 Overall sample size considerations

In order to achieve 90% power both for the primary analysis (PTA4 and SNR, Investigational Device vs. unaided) and the primary safety analysis, 50 evaluable subjects are needed. Each arm SSD and Conductive/Mixed should at least consist of 13 patients to assure a power of 90% in both arms for the primary analyses.

#### 2 STUDY POPULATIONS

#### 2.1 Definition of Study Populations

The final definition of the analysis sets (ITT, PP and Safety) will be taken at the clean file meeting before database lock.

| STATISTISKA KONSULTGRUPPEN | N Statistical Analysis Plan |
|---|---|

#### 2.1.1 Intent-to-Treat Population (Full Analysis Set)

The Intention-to-Treat population (ITT) will include all subjects who have undergone surgical intervention.

#### 2.1.2 Per-Protocol Population

The Per Protocol population (PP) will include subjects that have completed the investigation according to the protocol. Subjects that were incorrectly included or were considered major protocol violators should be removed from the PP population.

#### 2.1.3 Safety Population

The Safety population consists of all surgically treated subjects

#### 3 STUDY VARIABLES

#### 3.1 Baseline variables

#### 3.1.1 Demographics

- Age (years), calculated from date of birth and date of
- Gender
- Ethnicity
- Nicotine use
- Site
- Country

#### 3.1.2 Baseline Characteristics

- Treatment ear
  - o Right
  - o Left
- Type of hearing loss
  - Conductive/mixed
  - o SSD
- Aetiology
  - o (Chronic) Infection
  - o Tumour
  - o Trauma
  - o Malformation
  - o Otosclerosis
  - o Other
- Current hearing aid
  - Yes
  - o No

#### 3.1.3 Medical and Surgical History

- Medical history will be coded using CTCAE.
- Surgical history will be coded using CTCAE.

| STATISTISKA KONSULTGRUPPEN | Statistical Analysis Plan |
|---|---|
| Clinical performance of a new implant system for bone | Protocol No:<br>CBAS5539 |

#### 3.1.4 Prior and Concomitant Medications

Prior medication is defined as medication used up surgery. Concomitant medications are medications used from Surgery to end of study. Medications are coded according to WHO CC ATC.

#### 3.1.5 Concomitant Treatments/Procedures

Concomitant Treatments/Procedures between Visit 1 and end of study will be collected. These terms will not be coded.

#### 3.2 Efficacy Variables/endpoints

#### 3.2.1 Primary Efficacy Variables/endpoints

- Threshold audiometry: PTA4 (mean of 500, 1000, 2000 and 4000Hz) at visit 1 (unaided) vs 3 months post-surgery (aided).
- Change in Adaptive speech recognition in noise (50% performance) from unaided versus Investigational device at the 3 months visit.

#### 3.2.2 Secondary Efficacy Variables/endpoints

- Abbreviated Profile of Hearing Aid Benefit (APHAB) at visit 1 (unaided), m 3, m 6 and m 12:
  - Global score
  - Ease of Communication
  - Reverberation
  - Background Noise
  - Aversiveness
- Thresholds audiometry: PTA-4, 250, 500, 1000, 2000, 3000, 4000, and 6000
   Hz at visit 1, w 4, m 3, m 6 and m 12
- Speech perception in quiet (50dB, 65dB and 80dB SPL) at visit 1, w 4, m 3, m 6 and m 12
- Adaptive speech recognition in noise (50% performance) at visit 1, w 4, m 3, m 6 and m 12
- Feedback measurement at each frequency at visit w 4, w 6, m 3, m 6 and m
   12
- Generic quality of life scale: Health Utility Index (HUI) at visit 1 (unaided), m 3, m 6 and m 12:
  - Health related quality of life score for overall health
  - Vision score
  - o Hearing score
  - Speech score
  - o Ambulation/mobility score
  - Dexterity score
  - o Self-care score
  - o Emotion score
  - Cognition score
- The Speech, Spatial and Qualities of Hearing Scale (SSQ) at visit 1 (unaided), m 3, m 6 and m 12

#### Surgical variables

- Soft tissue thickness (mm)
- Surgery time (time of first incision to time of last suture), (min)

| STATISTISKA KONSULTGRUPPEN | Statistical Analysis Plan | |
|---|---|---|
| Clinical performance of a new implant system for bone | Protocol No CBAS5 | |
| conduction hearing | Version: 1.0 | Page 12 of |

- Type of anaethesia
- Soft tissue thinning performed
  - o Yes
  - o No
- Bone polishing/removal below the actuator site performed
- BI300 length
  - o 3 mm
  - o 4 mm
- Location of BI300 Implant
- Surgical incision/location

Questions about usage will be collected at w 6, w 12, m 6 and m 12:

- Daily use of sound processor (hours/day)
- Softpad use
- Question about comfort with the SP, using VAS, will be collected at w 4, w 6, m 3, m 6 and m 12.
- Magnet choice will be recorded at w 4, w 6, w 12, m 6 and m 12.

BC Direct thresholds at visit 1, w 4, w 6, m 3, m 6 and m 12

#### 3.3 Safety Variables/Endpoints

#### 3.3.1 Implant site evaluation

Evaluation about numbness around the implant site will be performed at w 2, w4, w 6, m 3, m 6 and m 12.

- Total sensibility %
- Gnostic sensibility % (cotton swab) at 30 mm and 60 mm for Cranial, Caudal, Anterior and Posterior
- Vital sensibility % (sharp wodden) at 30 mm and 60 mm for Cranial, Caudal, Anterior and Posterior

## 3.3.2 Adverse Events

Adverse events from visit 2 and onward will be presented.

- Adverse Event (AE) is all reported events
- Adverse Device Effect (ADE) is events that is Related to the device (Probably) or Related to the procedure (Probably)
- Serious Adverse Event (SAE) is events that has been marked as Serious
- Serious Adverse Device Effect (SADE) is events that has been marked as Serious and also marked as Related to the device (Probably) or Related to the procedure (Probably)
- The following AEs are defined as adverse events of special interest (AESIs):
  - o AE that interfere with the daily use of the medical device(s)
  - AE at the site of the implant that lead to
    - Revision surgery including explantation
    - Severe soft tissue complication
    - Prescription of antibiotics

#### 3.3.3 Device deficiency

Device deficiency will be collected at d 0, w 2, w 4, w 6, m 3, m 6 and m 12.

- Has any device deficiency occurred?
  - o Yes

| STATISTISKA KONSULTGRUPPEN | Statistical Analysis Plan |
|---|---|
| Protocol: Clinical performance of a new implant system for bone | Protocol No CBAS |

o No

#### 3.3.4 Audiogram

Audiogram at Visit 1, Air condition/Bone conduction, Right/Left (transferred to test side/Non test side), Unmasked/Masked for 250, 500, 750, 1000, 1500, 2000, 3000, 4000, 6000 and 8000 Hz. At 3 months visit and 12 months visit test side audiogram, bone conduction (unmasked and if needed masked) thresholds at 250, 500, 750, 1000, 1500, 2000, 3000, 4000 and 6000Hz will be collected.

#### 4 STATISTICAL METHODOLOGY

# 4.1 General Methodology

Since all included subjects will have measurements of the primary and important secondary efficacy variables for unaided hearing, with the Investigational device and with a Baha power sound processor on a Baha Softband, all statistical analyses will be paired. All statistical analyses will be non-parametric. In order to choose the most powerful test, the Fisher's non-parametric permutation test for paired observations will be used for all paired analyses of continuous variables. The permutation tests use the measured values and not only the ranks in the calculations. For paired analysis of dichotomous and ordered categorical variables the Sign test will be used.

The analyses will be performed in the following priority:

- 1. Investigational Device vs. Unaided
- 2. Investigational Device vs. Baha power sound processor on a Baha Softband

In addition to the change variables the distribution of all efficacy variables will be presented by visit, where applicable.

The main efficacy analysis will be performed on the ITT population and complementary efficacy analyses will be performed on the PP population. The main analysis will be performed after the 3 month visit. A complementary analysis will be performed 9 months after the main analysis (12-month visit). All significance tests will be one-sided and performed at the 2.5% significance level to demonstrate an improvement with Investigational Device.

The hierarchical testing procedure below is introduced to guarantee that the probability of Type I error is < 2.5% for all confirmative statements. The order of the hierarchical testing procedure will be:

- 1. PTA 4 pre-operative unaided vs 3 months (Primary efficacy analysis)
- 2. Adaptive speech recognition in noise (50% performance), speech to noise ratio (SNR) pre-operative unaided vs 3 months
- 3. Speech in quiet at 65dB SPL pre-operative unaided vs 3 months
- 4. APHAB Global pre-operative unaided vs 3 months aided
- 5. Hearing attribute (HUI-III) pre-operative unaided vs 3 months
- 6. Mean of the 12 items in the SSQ pre-op unaided vs 3 months

If the first analysis is significant the probability mass 0.025 will go to the second analysis. If the second analysis is also significant the probability mass 0.025 will go to the third analysis and so on. When the first non-significant analysis is reached this and all analyses thereafter will be non-confirmative while the previous analyses will be confirmative. If the first analysis is non-significant no analysis will be confirmative.

| STATISTISKA KONSULTGRUPPEN | Statistical Analysis Plan |
|---|---|
| Clinical performance of a new implant system for bone | Protocol No:<br>CBAS5539 |

The hierarchical testing will be made for each arm separately (SSD and Mixed/Conductive) and not totally.

We plan to analyse the similarity of the primary efficacy results among sites using non-parametric one way analyses of variance (Kruskal-Wallis test) of the difference between Unaided and ATB at 3 months. This will only be made totally and not by SSD and Mixed conductive.

Imputation of missing values will be performed for all efficacy variables. No imputation of baseline values or baseline carry forward will be made. Imputations will be made according to the following rules:

- If a value is missing at the end of a patient, last observation will be carried forward.
- 2. If a missing value is occurring between two time points with values, an interpolation will be made for continuous variables and for categorical variables the value from the previous visit will be carried forward.

The distribution of continuous variables as well as change in continuous variables will be given as n, mean, SD, SEM, Median, Min and Max and the distribution of dichotomous and categorical variables will be given as number and percentages. One sided 97.5% CI will be presented where applicable.

Numbness, Adverse Events, Device deficiencies, Comfort, Usage, Surgical variables, Demographics, Baseline, Questions, Magnet strength variables will only be analysed descriptively.

#### 4.2 Timing of analyses

The main efficacy analysis is made at 3 months and another follow-up analysis at 12 months. The primary Safety analysis will be made at 6 months.

- When locking the data at 3 months both efficacy and safety will be evaluated.
- When locking the data at 6 months only safety will be evaluated.
- When locking the data at 12 months both efficacy and safety will be evaluated.

#### 4.3 Patient Disposition and Data Sets Analysed

The number of subjects included in each of the ITT, PP and Safety populations will be summarised. Subjects who completed the study and subjects who withdrew from study prematurely will also be presented with a breakdown of the reasons for withdrawal by treatment group for the ITT, PP and safety populations.

#### 4.4 Protocol Deviations

Major protocol deviations are those that are considered to have an effect on the analysis. The number of patients with major protocol deviations will be summarised per treatment group. A list of protocol deviations will be produced.

# 4.5 Demographics and Baseline Characteristics

Demographics and baseline characteristics will be descriptively summarised by SSD and Mixed/Conductive and totally for the ITT and PP populations.

| STATISTISKA KONSULTGRUPPEN | Statistical Analysis Plan |
|---|---|
| Protocol: Clinical performance of a new implant system for bone | Protocol No:<br>CBAS5 |

#### 4.6 Pre operation variables

Pre operation variables will be summarised by SSD and Mixed/Conductive and totally for the ITT and PP populations and analysed according to the methods described in section "General Methodology" above.

## 4.7 Medical and Surgical History

Medical and surgical history, one at a time, will be summarised by CTCAE term by SSD and Mixed/Conductive and totally for ITT population.

#### 4.8 Prior and Concomitant Medications

Prior and concomitant medication will be summarised by higher level anatomical therapeutic classification (ATC) group and generic term by SSD and Mixed/Conductive and totally for ITT population.

#### 4.9 Concomitant Treatments/Procedures

Concomitant treatments/procedures will be listed for the ITT population. A special mark-up will be done whether to tell if the treatment was performed before or/after surgery.

## 4.10 Efficacy Analyses

#### 4.10.1 Primary Efficacy Analysis

Primary efficacy analysis will be determined by analysis of change in free-field threshold audiometry: PTA4 (mean of 500, 1000, 2000 and 4000Hz) and change in Adaptive speech recognition in noise (50% performance), from unaided versus Investigational device at the 3 months visit for the ITT population, using Fisher's one-sided non-parametric permutation test for paired observations at a significance level of 0.025 to demonstrate an improvement in PTA4. Each arm SSD and Conductive/Mixed will be tested separately. Both PTA4 and SIQ must be significant at alpha 0.025 for the primary analysis to be considered as confirmative in each arm separately. In addition, a pooled analysis for all subjects will be made.

Group mean free-field PTA4 (average of 500, 1000, 2000, and 4000 Hz) with the Osia System at the 3-month postoperative interval will be improved over that measured preoperatively in the unaided condition (baseline).

This endpoint is represented by the following hypotheses:

$$H_0: \mu_F - \alpha_0 \ge 0,$$

$$H_a$$
:  $\mu_F - \alpha_0 < 0$ ,

where:

 $\alpha_0$  = baseline preoperative PTA4;

 $\mu_F$  = mean follow-up PTA4 3 months postoperative.

Group mean Adaptive speech recognition in noise (50% performance), speech to noise ratio (SNR) with the Osia System at the 3-month postoperative interval will be improved over that measured preoperatively in the unaided condition.

| STATISTISKA KONSULTGRUPPEN | Statistical | Statistical Analysis Plan |
|---|---|---|

This endpoint is represented by the following hypotheses:

$$H_0: \mu_F - \alpha_0 \ge 0$$
,

$$H_a$$
:  $\mu_F - \alpha_0 < 0$ ,

where:

 $\alpha_0$  = baseline preoperative Adaptive speech recognition in noise (50% performance), speech to noise ratio (SNR);

 $\mu_F$  = mean follow-up Adaptive speech recognition in noise (50% performance), speech to noise ratio (SNR) 3 months postoperative.

A sensitivity analysis of the primary variable will be done for complete cases.

The primary analyses will be performed regardless of what Osia Fitting Software version (1.0.2 OFS or 1.0.3 OFS) used at 3 months (see chapter 4.12).

#### 4.10.2 Secondary Efficacy Analyses

The secondary efficacy objectives in the hierarchical testing will be tested using the following hypothesis:

Group mean Speech in quiet at 65dB with the Osia System at the 3-month postoperative interval will be improved over that measured preoperatively in the unaided condition.

This endpoint is represented by the following hypotheses:

$$H_0: \mu_F - \alpha_0 \le 0$$
,

$$H_a: \mu_F - \alpha_0 > 0$$
,

where:

 $\alpha_0$  = baseline preoperative word recognition score;

 $\mu_F$ = mean follow-up word recognition score 3 months postoperative.

Group mean APHAB Global score with the Osia System at the 3-month postoperative interval will be improved over that measured preoperatively in the unaided condition.

This endpoint is represented by the following hypotheses:

$$H_0: \mu_F - \alpha_0 \ge 0$$
,

$$H_a$$
:  $\mu_F - \alpha_0 < 0$ ,

where:

 $\alpha_0$  = baseline preoperative APHAB Global score;

 $\mu_F$ = mean follow-up APHAB Global score 3 months postoperative.

| STATISTISKA KONSULTGRUPPEN | Statistica | l Analysis Plan |
|---|---|---|

Group mean Hearing attribute (HUI-III) with the Osia System at the 3-month postoperative interval will be improved over the preoperative hearing situation.

This endpoint is represented by the following hypotheses:

$$H_0: \mu_F - \alpha_0 \le 0$$
,

$$H_a: \mu_F - \alpha_0 > 0$$
,

where:

 $\alpha_0$  = baseline preoperative Hearing attribute (HUI-III);

 $\mu_F$ = mean follow-up Hearing attribute (HUI-III) 3 months postoperative.

Group mean of the 12 items in the SSQ with the Osia System at the 3-month postoperative interval will be improved over the preoperative hearing situation.

This endpoint is represented by the following hypotheses:

$$H_0$$
:  $\mu_F - \alpha_0 \leq 0$ ,

$$H_a$$
:  $\mu_F - \alpha_0 > 0$ ,

where:

 $\alpha_0$  = baseline preoperative mean of the 12 items in the SSQ;

 $\mu_F$ = mean follow-up mean of the 12 items in the SSQ 3 months postoperative.

Comparison regarding change from unaided hearing (if applicable) to Investigational device will be done according to the general methodology with Fisher's non-parametric permutation test for paired observations for the following variables:

- APHAB at 3, 6 and 12 months
- Threshold audiometry: PTA4 (Mean of 500, 1000, 2000 and 4000 Hz) at 4 weeks, 6 and 12 months
- Threshold audiometry: 250, 500, 1000, 2000, 3000, 4000 and 6000 Hz at 4 weeks, 3, 6, and 12 months
- Adaptive speech recognition in noise (50% performance) at 4 weeks, 3, 6 and 12 months
- Speech in quiet (50dB, 65dB and 80dB) at 4 weeks, 3, 6 and 12 months
- Feedback measurement at each frequency at 4 and 6 weeks, 3, 6 and 12 months
- HUI-III at 3, 6 and 12 months
- SSQ at 3, 6 and 12 months

Comparison of the Investigational device with a Baha Power sound processor worn on a Baha Softband will be done according to the general methodology with Fisher's non-parametric permutation test for paired observations for the following variables:

- Threshold audiometry: PTA4 (Mean of 500, 1000, 2000 and 4000 Hz) at 4 weeks, 3, 6 and 12 months
- Threshold audiometry: 250, 500, 1000, 2000, 3000, 4000 and 6000 Hz at 4 weeks, 3, 6, and 12 months

| STATISTISKA KONSULTGRUPPEN | Statistica | l Analysis Plan |
|---|---|---|

- Adaptive speech recognition in noise (50% performance) at 4 weeks, 3, 6 and 12 months
- Speech in quiet (50dB, 65dB and 80dB) at 4 weeks, 3, 6 and 12 months
- BC Direct at 4 and 6 weeks, 3, 6 and 12 months.

Choice of SP magnet and change of SP magnet. Changes in SP magnet strength will also be presented graphically in a flow graph.

All secondary efficacy analyses will be performed for both the ITT population and PP population. PTA4 will also be analysed for the PP population in the same fashion as in the primary analysis.

Analyses of Threshold Audiometry, Adaptive speech recognition in noise and Speech in quiet, BC Direct, HUI, APHAB and SSQ will be made totally and also by SSD and Conductive/Mixed patients. This will be made only for the ITT population.

#### 4.10.3 Tertiary Efficacy Analyses

As tertiary efficacy analysis adaptive speech in noise [speech-to-noise ratio, 50% speech understanding] with a current hearing aid (if used by the patient) will be presented. Summarization will be made for the ITT population totally and by SSD and Mixed/Conductive (if sufficient data is collected).

## 4.11 Safety Analyses

The primary safety analysis will be evaluated at 6 months.

#### 4.11.1 Implant site evaluation

Evaluation about numbness will be presented by visit. Changes from first measurement may be evaluated.

# 4.11.2 Adverse Events

AEs will be included in the summaries for safety population.

A summary of subjects reporting at least one of the following AEs will be presented in an overview table:

- Any AE
- Any SAE
- Any Adverse Device Effect (ADE)
- Any Serious Adverse Device Effect (SADE)
- Any AESI

Summaries by CTCAE term presenting n (%) of AEs and n (%) of subjects with at least one AE will be provided for:

- All AE
- All SAE
- All Adverse Device Effect (ADE)
- All Serious Adverse Device Effect (SADE)
- All AESI

#### 4.11.3 Device deficiency

Device deficiency will be presented by visit.

| STATISTISKA KONSULTGRUPPEN | Statistica | l Analysis Plan |
|---|---|---|

#### 4.11.4 Audiogram

Audiogram (Air and Bone conduction), test side for 250, 500, 750, 1000, 1500, 2000, 3000, 4000, 6000 and 8000 Hz by SSD and Conductive/Mixed patients will be presented at visit 1, 6 and 8. At visit 6 and 8 is only bone conduction performed.

# 4.12 Handling of change in Osia version of Fitting Software

Due to the change in version of Osia Fitting Software (OFS) during the study (from 1.0.2 to 1.0.3) analyses are planned for taking care of this. All patients that are already fitted with OFS version 1.0.2 will switch from 1.0.2 OFS to the new 1.0.3 OFS at a certain visit (1 year at the latest) and some will use the new 1.0.3 OFS from start. This means that some patients will, at a certain time point, have done their measurements based on different OFS. We do not intend to change the primary efficacy analyses due to the change in OFS.

When both 1.0.2 OFS and 1.0.3 OFS are measured (at a certain visit when the change is implemented) the new 1.0.3 OFS version will be used in the planned analyses.

The following analyses are planned due the change of OFS:

- 1. Frequency of "OFS change visit" in order to present the distribution of when the change took place. If a patient used the 1.0.3 from the beginning Visit 4 Fitting will be presented.
- 2. Descriptives and changes from unaided for free-field thresholds, speech in quiet test and speech in noise test by visit will be presented by 1.0.2 OFS and 1.0.3 OFS without statistically testing.
- 3. For the patients who initially used 1.0.2 OFS the free-field thresholds, the speech in quiet test and the speech in noise test will be compared at the visit when the change took place. Results will be summarized for 1.0.2 OFS, 1.0.3 OFS and for the difference between the versions. This will be made totally but also by visit (when the change took place). Scatter plots of 1.0.2 OFS (x) vs 1.0.3 OFS (y) with visit where the change took place as group (colour/symbol) indicator will be produced. In addition, line plots of measure (y) vs OFS version (y), one line per patient with visit where the change took place as group (colour/symbol) indicator will be produced.

#### 5 INTERIM ANALYSES

An interim safety analysis will be performed when all subjects at the site in Melbourne have completed the 3 month visit (i.e. visit 6). Based on the result of this interim analysis a 'go/no go' decision will be taken if to proceed with the investigation at the other sites. Focus of this safety analysis will be on reported Serious Adverse Event (SAEs) and Adverse Event of Special Interest (AESIs), i.e.:

- AE that interfere with the daily use of the medical device(s)
- AE at the site of the implant that lead to
  - Revision surgery including explantation
  - Severe soft tissue complication
  - o Prescription of antibiotics

| STATISTISKA KONSULTGRUPPEN | Statistical | Analysis Plan |
|---|---|---|

The 'go/no go' decision will be taken by the co-ordinating investigator and the Sponsor in collaboration with the principal investigator at the Melbourne site

# 6 CHANGES OF ANALYSIS FROM PROTOCOL

No changes of the analyses according to the protocol are made.

# 7 LISTING OF TABLE, FIGURES AND LISTINGS

# 7.1 Listing of Tables

| Table 14.1.1<br>Table 14.1.2 | Patient Disposition and Data Sets Analysed<br>Protocol Deviations Leading to Exclusion from PP Population (ITT<br>Population) |
|---|---|
| Table 14.1.3.1<br>Table 14.1.3.2<br>Table 14.1.4.1 | Demographics and Baseline Characteristics (ITT Population) Demographics and Baseline Characteristics (PP Population) Pre operation (ITT Population) |
| Table 14.1.4.2 | Pre operation (PP Population) |
| Table 14.1.5.1 | Audiogram (air) at visit 1, 6 and 8 - SSD patients (Safety Population) |
| Table 14.1.5.2 | Audiogram (bone) at visit 1, 6 and 8 - SSD patients (Safety Population) |
| Table 14.1.5.3 | Audiogram (air) at visit 1, 6 and 8 - conductive patients (Safety Population) |
| Table 14.1.5.4 | Audiogram (bone) at visit 1, 6 and 8 - conductive patients (Safety Population) |
| Table 14.1.6 | Medical History (ITT Population) |
| Table 14.1.7 | Surgical History (ITT Population) |
| Table 14.1.8.1 | Prior Medications (ITT population) |
| Table 14.1.8.2 | Concomitant Medications (ITT population) |
| Table 14.1.9 | Listing of Concomitant Treatments/Procedures (ITT population) |
| Table 14.2.1.1 | Threshold Audiometry - Free field ATB System vs Unaided (ITT Population) |
| Table 14.2.1.2 | Threshold Audiometry - Free field ATB System vs Unaided (PP Population) |
| Table 14.2.2.1 | Adaptive speech recognition in noise and Speech in quiet ATB |
| T-bl- 44 0 0 0 | System vs Unaided (ITT Population) |
| Table 14.2.2.2 | Adaptive speech recognition in noise and Speech in quiet ATB vs Unaided (PP Population) |
| Table 14.2.3.1 | BC Direct (ITT Population) |
| Table 14.2.3.2 | BC Direct (PP Population) |
| Table 14.2.4.1 | HUI (ITT Population) |
| Table 14.2.4.2 | HUI (PP Population) |
| Table 14.2.5.1 | APHAB (ITT Population) |
| Table 14.2.5.2 | APHAB (PP Population) |
| Table 14.2.6.1 | The Speech, Spatial and Qualities of Hearing Scale (SSQ) (ITT Population) |
| Table 14.2.6.2 | The Speech, Spatial and Qualities of Hearing Scale (SSQ) (PP Population) |
| Table 14.2.7.1 | Surgery (ITT population) |
| Table 14.2.7.2 | Surgery (PP population) |
| Table 14.2.8.1 | Magnet strength (ITT population) |
| Table 14.2.8.2 | Magnet strength (PP population) |
| Table 14.2.9.1 | Daily use and soft-pad use (ITT population) |

| STATISTISKA KONSULTGRUPPEN | Statistica | l Analysis Plan |
|---|---|---|

| Table 14.2.9.2<br>Table 14.2.10.1 | Daily use and soft-pad use (PP population) Threshold Audiometry - Free field ATB System vs Unaided (SSD |
|---|---|
| - | patients ITT Population) |
| Table 14.2.10.2 | Adaptive speech recognition in noise and Speech in quiet ATB System vs Unaided (SSD patients ITT Population) |
| Table 14.2.10.3 | BC Direct (SSD patients ITT Population) |
| Table 14.2.10.4 | HUI (SSD patients ITT Population) |
| Table 14.2.10.5 | APHAB (SSD patients ITT Population) |
| Table 14.2.10.6 | The Speech, Spatial and Qualities of Hearing Scale (SSQ) (SSD patients ITT Population) |
| Table 14.2.11.1 | Threshold Audiometry - Free field ATB System vs Unaided (Conductive/Mixed patients ITT Population) |
| Table 14.2.11.2 | Adaptive speech recognition in noise and Speech in quiet ATB System vs Unaided (Conductive/Mixed patients ITT Population) |
| Table 14.2.11.3 | BC Direct (Conductive/Mixed patients ITT Population) |
| Table 14.2.11.4 | HUI (Conductive/Mixed patients ITT Population) |
| Table 14.2.11.5 | APHAB (Conductive/Mixed patients ITT Population) |
| Table 14.2.11.6 | The Speech, Spatial and Qualities of Hearing Scale (SSQ) |
| | (Conductive/Mixed patients ITT Population) |
| Table 14.2.12.1 | Threshold Audiometry - Free field ATB System vs Softband (ITT |
| | Population) |
| Table 14.2.12.2 | Threshold Audiometry - Free field ATB System vs Softband (PP Population) |
| Table 14.2.12.3 | Threshold Audiometry - Free field ATB System vs Softband (Conductive/Mixed patients ITT Population) |
| Table 14.2.12.4 | Threshold Audiometry - Free field ATB System vs Softband (SSD patients ITT Population) |
| Table 14.2.13.1 | Adaptive speech recognition in noise and Speech in quiet ATB System vs Softband (ITT Population) |
| Table 14.2.13.2 | Adaptive speech recognition in noise and Speech in quiet ATB System vs Softband (PP Population) |
| Table 14.2.13.3 | Adaptive speech recognition in noise and Speech in quiet ATB System vs Softband (SSD patients ITT Population) |
| Table 14.2.13.4 | Adaptive speech recognition in noise and Speech in quiet ATB System vs Softband (Conductive/Mixed patients ITT Population) |
| Table 14.3.1.1 | Summary of Adverse Events (Safety Population) |
| Table 14.3.1.2 | Adverse Events (AE), by CTCAE Term (Safety Population) |
| Table 14.3.1.3 | Adverse Device Events (ADE), by CTCAE Term (Safety Population) |
| Table 14.3.1.4 | Serious Adverse Events (SAE), by CTCAE Term (Safety |
| | Population) |
| Table 14.3.1.5 | Serious Adverse Device Events (SADE), by CTCAE Term (Safety Population) |
| Table 14.3.2 | Pain and Numbness (Safety Population) |
| Table 14.3.3 | Device deficiency (Safety Population) |

# 7.2 Listing of Figures

To be decided later.

# 7.3 Listing of Listings

Listings are decided outside of this SAP.

| STATISTISKA KONSULTGRUPPEN | Statistical Analysis Plan |
|---|---|
| conduction hearing | Version:<br>1.0 Page 22 of<br>22 |

# 8 REFERENCES

# 9 APPENDIX